CLINICAL TRIAL: NCT05372887
Title: A Phase 2, Double-Blind, Randomized, Multicenter, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Daily Bedtime TNX-102 SL in Participants With PTSD
Brief Title: Safety and Efficacy Study of TNX-102 SL in Participants With PTSD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to business reasons.
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNX-CY-P308
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TNX-102 SL, 5.6 mg (Experimental): 2 x TNX-102 SL, 2.8 mg Tablets taken sublingually each day at bedtime for 12 weeks.
  Interventions: Drug: TNX-102 SL
- Placebo (Placebo Comparator): 2 x Placebo Tablet taken sublingually each day at bedtime for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TNX-102 SL — Patients will take 2 tablets of randomly assigned study drug sublingually each day at bedtime starting on Day 1 for 12 weeks
  Other Names: Low dose cyclobenzaprine sublingual tablets
  Arms: TNX-102 SL, 5.6 mg
Drug: Placebo — Patients will take 2 tablets of randomly assigned study drug sublingually each day at bedtime starting on Day 1 for 12 weeks
  Other Names: Placebo sublingual tablets
  Arms: Placebo

SUMMARY:
This is a 12-week, multicenter, randomized, double-blind, placebo-controlled, fixed-dose study that will investigate the efficacy and safety of 5.6 mg TNX-102 SL (2 x 2.8 mg tablets)-a sublingual formulation of cyclobenzaprine. Following successful screening and randomization, eligible patients will have a telephonic visit at week 2 and then return regularly to the study clinic for monthly visits for assessments of efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 75 years of age, at the time of signing ICF, inclusive.
* Diagnosed with current (past month) PTSD as determined by the MINI 7.0.2 Module H (PTSD).
* Index trauma(s) resulting in PTSD must meet DSM-5 Criterion A for PTSD as described in the CAPS 5, must have occurred within 9 years of Screening Visit 1, and must have occurred when the participant was ≥18 years of age.
* Willing and able to withdraw and refrain from opioids for the course of the study.
* Willing to refrain from use of all other formulations of cyclobenzaprine for the course of the study.
* Willing and able to refrain from antidepressants and other excluded medications.
* Capable of reading and understanding English and able to provide written informed consent to participate.
* Willing to comply with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.
* If female, either not of childbearing potential or practicing a medically acceptable method of birth control throughout the study.
* Body mass index (BMI) within the range 17.5 - 35 kg/m^2 (inclusive).

Exclusion Criteria:

* Current or ongoing exposure to the trauma that resulted in the PTSD (ie, non-work-related trauma such as ongoing domestic abuse).
* Increased risk of suicide, based on the investigator's judgment that is of a severity that is not appropriate for outpatient management, or that warrants additional therapy excluded by the protocol.
* Significant (eg, moderate or severe) comorbid traumatic brain injury (TBI) by history.
* Severe depressive symptoms at screening or baseline.
* Clinically significant laboratory abnormalities based on screening laboratory tests and/or medical history in the investigator's opinion.
* Use of antidepressant medication within 2 months of baseline.
* Female participants who are pregnant or lactating.
* History of serotonin syndrome, severe allergic reaction or bronchospasm or known hypersensitivity to cyclobenzaprine or the excipients in TNX-102 SL or placebo formulations.
* Seizure disorder.
* Current moderate or severe sleep apnea not well controlled by positive airway pressure (PAP) or oral (mouthpiece) devices.
* Has received any other investigational drug within 90 days before Screening or has taken cyclobenzaprine within 21 days of the Randomization visit.
* Previous participation in any other study with TNX-102 SL.
* Family member of investigative staff.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in the total Clinician Administered PTSD Scale (CAPS-5) for DSM-5 at Week 12. | Day 1, Week 4, Week 12
  To evaluate the efficacy of the TNX-102 SL (cyclobenzaprine HCl sublingual tablets) using the Clinician Administered PTSD Scale for Diagnostic and Statistical Manual of Mental Disorders, fifth edition (CAPS-5) total symptom severity score in a 12-week study.

SECONDARY OUTCOMES:
Clinical Global Impression - Severity change from Baseline to Week 12 | Day 1, Week 4, Week 8, Week 12
  CGI-S to assess global severity change from baseline to Week 12
Change from baseline in the disruption of psychosocial functioning assessed using the Sheehan Disability Scale (SDS) after 12 weeks of treatment. | Day 1, Week 4, Week 8, Week 12
  SDS to assess psychosocial functioning change from baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sullivan, MD, Study Director — Tonix Pharmaceuticals
Locations (3):
- Kenya (3):
  - Aga Khan University Clinical Research Unit, Nairobi
  - Centre for Clinical Research at KEMRI-Nairobi, Nairobi
  - Moi University Clinical Research Centre, Nairobi

IPD SHARING:
Plan to Share IPD: Undecided